CLINICAL TRIAL: NCT02464124
Title: A Randomized, Double-blind, Controlled Trial Comparing Nitazoxanide Plus Lactulose With Lactulose Alone Treatment of Overt Hepatic Encephalopathy
Brief Title: Nitazoxanide Plus Lactulose Versus Lactulose Alone Treatment of Hepatic Encephalopathy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, sponsor investigator, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hepatic encephalopathy
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Encephalopathy, Hepatic
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — nitazoxanide; Lactulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lactulose plus nitazoxanide (Experimental): * Nitazoxanide dosing: 500 mg tablets twice daily
  * Lactulose dosing: 30-60 mL PO TID with goal 2-3 semisoft stools per day
  Interventions: Drug: Nitazoxanide; Drug: Lactulose
- Lactulose alone (Active Comparator): Lactulose dosing: 30-60 mL PO TID with goal 2-3 semisoft stools per day
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: Nitazoxanide — • Nitazoxanide dosing: 500 mg tablets twice daily
  Other Names: Alenia, Nitclean, Parazoxanide
  Arms: lactulose plus nitazoxanide
Drug: Lactulose — • Lactulose dosing: 30-60 mL PO TID with goal 2-3 semisoft stools per day
  Other Names: Laxolac, Duphlac

SUMMARY:
Hepatic encephalopathy (HE) is a reversible neuropsychiatric syndrome associated with chronic and acute liver dysfunction. It is characterized by cognitive and motor deficits of varying severity.

Treatment options include lactulose administered orally or by nasogastric tube or enema, non-absorbable antibiotics, and protein-restricted diets.

Nitazoxanide is an oral agent indicated for the treatment of infectious diarrhea caused by Crytpsporidiumparvum and Giardia lamblia. Basu and colleagues presented a pilot prospective study at the 2008 American Association for the Study of Liver Diseases meeting showing clinical improvement in HE among cirrhotic patients who received nitazoxanide and lactulose.

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) is a reversible neuropsychiatric syndrome associated with chronic and acute liver dysfunction. It is characterized by cognitive and motor deficits of varying severity.

Hepatic encephalopathy is caused by accumulation of nitrogenous substances, primarily ammonia, in the blood. In advanced stages it is referred to as hepatic coma which may be preceded by seizures. The treatment goal is to reduce nitrogen load from the GI tract and to improve central nervous system (CNS) status.

Treatment options include lactulose administered orally or by nasogastric tube or enema, non-absorbable antibiotics, and protein-restricted diets.

Lactulose is nonabsorbable disaccharides that are currently used as first line agents for the treatment of HE. Its action is thought to beconversion to lactic acid and acetic acid resulting in acidification of the gut lumen. This favors conversion of ammonia (NH3) to ammonium (NH4+), which is relatively membrane impermeable, and inhibits ammoniagenic coliform bacteria.

Nitazoxanide is an oral agent indicated for the treatment of infectious diarrhea caused by Crytpsporidiumparvum and Giardia lamblia. Basu and colleagues presented a pilot prospective study at the 2008 American Association for the Study of Liver Diseases meeting showing clinical improvement in HE among cirrhotic patients who received nitazoxanide and lactulose.

Mantry and colleagues showed that the number of hospitalizations and the duration of hospital stays were shortened for patients receiving combination therapy compared with those receiving lactulose monotherapy.

ELIGIBILITY:
Inclusion Criteria:

Age 18-70 years

Cirrhosis, defined by a combination of any of the following:

* Laboratory findings
* Endoscopic results
* Ultrasound
* Histology Overt hepatic encephalopathy

Exclusion Criteria:

* • Creatinine>1.5 mg/dl

  * Alcohol use within prior 4 weeks
  * Non-hepatic metabolic encephalopathy
  * Hepatocellular carcinoma
  * Degenerative CNS disease
  * Any significant psychiatric illness or other medical comorbidity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with total reversal of hepatic encephalopathy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Asem Elfert, Prof, Principal Investigator — hepatology dept-Tanta; Sherief Abd-Elsalam, lecturer, Study Director — hepatology dept-Tanta; Samah Soliman, lecturer, Study Chair — hepatology dept-Tanta; Walaa elkhalawany, lecturer, Study Chair — hepatology dept-Tanta; Rehab elsheshtawi, lecturer, Study Chair — hepatology dept-Tanta; Mennat-Allah Elsawaf, lecturer, Study Chair — hepatology dept-Tanta
Locations (1):
- Tanta university - faculty of medicine, Tanta, Elgharbia, Egypt